CLINICAL TRIAL: NCT02037126
Title: Psilocybin-facilitated Treatment for Cocaine Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Peter Hendricks, University Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND_121000
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Psilocybin; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Independent statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin administration (Experimental): Psilocybin will be administered in pill form at a dose of .36 mg/kg. Psilocybin will be administered in one session over the course of 8 hours.
  Interventions: Drug: Psilocybin
- Diphenhydramine administration (Active Comparator): Diphenhydramine will be administered in pill form at a dose of 100 mg. Diphenhydramine will be administered in one session over the course of 8 hours.
  Interventions: Drug: Diphenhydramine

INTERVENTIONS:
Drug: Psilocybin — this has been used in treating obsessive-compulsive disorders, cluster headaches, anxiety, and drug dependence.
  Other Names: psychedelic compound
  Arms: Psilocybin administration
Drug: Diphenhydramine — This drug will be used as the control. Diphenhydramine is a histamine blocker.
  Other Names: Benadryl
  Arms: Diphenhydramine administration

SUMMARY:
The primary purpose of this study is to evaluate the feasibility and estimate the efficacy of psilocybin-facilitated treatment for cocaine use. We also will monitor the impact of psilocybin-facilitated treatment on the use of other drugs and outcomes relevant to cocaine involvement.

MRI assessment is a unique aspect of this study. As a potential biological mechanism of psilocybin's effect includes changes in default mode network functional connectivity (Carhart-Harris et al., 2012), we will determine if psilocybin's therapeutic effects are mediated by such changes. Moreover, as Glx (a brain metabolite that reflects glutamate) abnormalities have been shown to play a role in cocaine addiction, we will determine if psilocybin impacts Glx in the anterior cingulate cortex and hippocampus.

DETAILED DESCRIPTION:
Individuals who are eligible to participate and provide informed consent will complete baseline questionnaires and be randomly assigned in a double-blind manner to the Psilocybin or Active Placebo group. The first MRI assessment will take place shortly thereafter using a 3T head-only Magnetic Resonance Imaging and Spectroscopy scanner (Magnetom Allegra, Siemens medial Solutions, Malvern, PA), optimized for neuroimaging applications.

Preparation sessions (see below) and the drug administration session will take place in a room at the Clinical Research Unit designed to be as comfortable, aesthetically pleasing (i.e., living-room like), and safe (e.g., no furniture with sharp corners or glass objects) as possible, with a directly adjacent, private restroom.

All participants will undergo four weekly preparation sessions of approximately 2 hours each. The purpose of these sessions is to: 1) develop strong therapeutic alliance between the participants and the primary therapist (Dr. Hendricks) and secondary therapist; 2) establish comfort and rapport between participants and the remainder of the research team; 3) discuss participants' aspirations with regard to their drug administration experience (e.g., What do participants hope to gain from their experience?); 4) discuss the treatment rationale and putative mechanisms of action of psilocybin; 5) obtain a detailed personal history of the participant, with a focus on those factors contributing to their current difficulties; 6) prepare participants for drug administration, including a detailed account of all potential effects of the drug; 7) discuss all aspects of the drug administration protocol (i.e., logistics and procedures), including plans of action in the event that participants experience acute distress; and 8) administer cognitive-behavioral treatment for cocaine use. Any participant who demonstrates significant anxiety, discomfort, or unease regarding drug administration at the conclusion of the four preparation sessions will be provided up to two additional preparation sessions. If these sessions are unsuccessful at mitigating the participant's anxiety, discomfort, or unease, the participant will be removed from the study.

Approximately one week after their final preparation session, participants will be instructed to eat a low-fat breakfast prior to presenting for their drug administration session at 8:00 am, approximately 1 hour before drug administration. A urine sample will be collected to verify drug-free status and participants will be encouraged to relax and reflect before drug administration. The drug administration session will take place over the course of 8 hours. The primary and secondary therapists will be present with participants throughout this session (at least one individual will always be present with the participant, even during brief intervals when one of the two therapists may be using the restroom). During this time, participants will be encouraged to lie down, use an eye mask to block external visual distraction, and use headphones through which a supportive music program will be played. Participants will be instructed to focus their attention on their inner experiences throughout the session.

Any participant reporting significant distress will be provided reassurance verbally or physically (e.g., with a supportive touch to the hand or shoulder). In the event that psychological distress is insufficiently managed with reassurance alone, medication will be administered under the guidance of the study physician.

Blood pressure will be assessed at regular intervals via automatic blood pressure monitor (e.g., pre-administration, and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-administration), and medication for the treatment of acute hypertension will be administered should blood pressure remain elevated at >200 systolic or >110 diastolic.

Seven hours after drug administration, when the major drug effects have subsided, participants will complete questionnaires assessing their experience. Participants will then be released into the care of a friend or family member (as arranged during preparation sessions) and instructed not to drive an automobile or engage in any other potentially dangerous activity for the remainder of the day. Participants will be provided with the primary therapist's pager number should they feel the need for support that evening.

Within 2 days after the drug administration session, participants will meet with the therapists for approximately 1 hour to discuss and reflect on their experience. The therapists will assess for potential adverse effects at this time. The second MRI session will take place shortly thereafter. Participants will then meet with the guide once per week over the next 4 weeks with an emphasis on integration of their medication session experience in the context of achieving abstinence from cocaine; continued cognitive-behavioral treatment for cocaine use will be provided during these follow-up meetings.

Long-term assessment visits will take place 3 and 6 months after the final therapy meeting. A battery of measures will be delivered at these times. At the conclusion of the 6-month assessment meeting, participants will be debriefed.

ELIGIBILITY:
Inclusion Criteria:

* 25 years of age and older
* Score of at least 3 on the Severity of Dependence Scale
* Desire to cease cocaine use as indicated by a goal of complete cocaine abstinence on the Thoughts about Abstinence questionnaire
* Ability to read/write in English
* No prior hallucinogen use or it will have been at least 3 years since their last use of a hallucinogen
* Availability of a friend or family member into whose care the participant can be released following their drug administration session.
* In good general health as assessed by detailed medical history and physical examination
* Abstinence from cocaine for at least 7 days prior to experimental drug administration as confirmed via urinalysis and no signs of intoxication on other drugs.

Exclusion Criteria:

* 24 years of age and younger
* Women who are pregnant or breast feeding
* Current psychiatric diagnoses other than substance abuse/dependence
* Current hypertension (exceeding 140 systolic and 90 diastolic at resting as described below)
* Use of tricyclic antidepressants, lithium, Selective Serotonin Reuptake Inhibitors, Monoamine Oxidase Inhibitors, haloperidol, St. John's Wort, or other antipsychotic medications, mood stabilizers, or medications with serotonin activity
* History of any psychotic disorders
* History of bipolar I or II disorder
* First or second-degree relatives with any psychotic disorders, or bipolar I or II disorders
* Current suicidal or homicidal ideation
* Planning to move from the Birmingham area in the next 6 months
* Contraindications of MRI (metallic objects in the body, claustrophobia, difficulty with prior MRI)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2024-05 (Actual); Study Completion 2024-05 (Actual)

PRIMARY OUTCOMES:
The difference between the psilocybin and placebo groups in the percentage of days abstinent from cocaine, verified by urine drug screen. | From the psilocybin or placebo administration session to end-of-treatment (approximately 4 weeks in most participants), from end-of-treatment to 12 weeks after end-of-treatment, and from 12 weeks after end-of-treatment to 24 weeks after end-of-treatment.
  Percentage of days abstinent from cocaine among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview and with biochemically verified cocaine presence as assessed via a urine drug screen.
The difference between the psilocybin and placebo groups in sustained/complete abstinence from cocaine, verified by urine drug screen. | From the psilocybin or placebo administration session to 24 weeks after end-of-treatment.
  Sustained/complete abstinence from cocaine among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview and with biochemically verified cocaine presence as assessed via a urine drug screen.
The difference between the psilocybin and placebo groups in time to cocaine lapse. | From the psilocybin or placebo administration session to 24 weeks after end-of-treatment.
  Number of days to first use of cocaine after the drug administration session among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview and with biochemically verified cocaine presence as assessed via a urine drug screen.

SECONDARY OUTCOMES:
The difference between the psilocybin and placebo groups in the severity of cocaine dependence. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Severity of Dependence Scale (SDS) among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in the severity of cocaine withdrawal symptoms. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Cocaine Selective Severity Assessment (CSSA) interview among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo).
The difference between the psilocybin and placebo groups in cocaine craving. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Cocaine Craving Questionnaire-Brief among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in situational cocaine abstinence self-efficacy. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Brief Situational Confidence Questionnaire among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in motivation to quit/remain abstinent, confidence in the ability to quit/remain abstinent, and perceived difficulty quitting/remaining abstinent. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Thoughts About Abstinence Questionnaire among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in depression, anxiety, and stress. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Depression, Anxiety, and Stress Scale (DASS-21) among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in satisfaction with life. | Within 48 hours after psilocybin or placebo administration, at end-of-treatment (approximately 4 weeks after psilocybin or placebo administration in most participants), at 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Ratings on the Satisfaction with Life Scale among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in income, employment, and living situation. | At 12 weeks after end-of-treatment, and at 24 weeks after end-of-treatment.
  Responses on a brief demographic questionnaire among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed via self-report.
The difference between the psilocybin and placebo groups in the percentage of days abstinent from alcohol. | From the psilocybin or placebo administration session to end-of-treatment (approximately 4 weeks in most participants), from end-of-treatment to 12 weeks after end-of-treatment, and from 12 weeks after end-of-treatment to 24 weeks after end-of-treatment.
  Percentage of days abstinent from alcohol among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview.
The difference between the psilocybin and placebo groups in the percentage of days abstinent from heavy alcohol use. | From the psilocybin or placebo administration session to end-of-treatment (approximately 4 weeks in most participants), from end-of-treatment to 12 weeks after end-of-treatment, and from 12 weeks after end-of-treatment to 24 weeks after end-of-treatment.
  Percentage of days abstinent from heavy alcohol use among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview.
The difference between the psilocybin and placebo groups in the percentage of days abstinent from tobacco. | From the psilocybin or placebo administration session to end-of-treatment (approximately 4 weeks in most participants), from end-of-treatment to 12 weeks after end-of-treatment, and from 12 weeks after end-of-treatment to 24 weeks after end-of-treatment.
  Percentage of days abstinent from tobacco among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview.
The difference between the psilocybin and placebo groups in the percentage of days abstinent from cannabis. | From the psilocybin or placebo administration session to end-of-treatment (approximately 4 weeks in most participants), from end-of-treatment to 12 weeks after end-of-treatment, and from 12 weeks after end-of-treatment to 24 weeks after end-of-treatment.
  Percentage of days abstinent from cannabis among subjects in each of the arms (subjects receiving psilocybin and subjects receiving placebo) assessed with the Timeline Followback Interview.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S. Hendricks, Ph.D., Principal Investigator — UAB Department of Psychiatry
Locations (1):
- UAB Outpatient Clinical Research Unit, Birmingham, Alabama, United States